CLINICAL TRIAL: NCT05430126
Title: Hepatotoxicity Related to Protein Kinase Inhibitors in Cancer Patients : an Observational and Retrospective Study Using the FDA Adverse Event Reporting System (FAERS)
Brief Title: Hepatotoxicity Related to Protein Kinase Inhibitors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Miao Yan, PhD, Associate Professor, Central South University
Other Study IDs: CSU20220619
Record Dates: First submitted 2022-06-19; First posted 2022-06-24 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Protein Kinase Inhibitors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Protein Kinase Inhibitor — This retrospective pharmacovigilance study will include protein kinase inhibitor and exclude those drugs known to cause hepatotoxicities

SUMMARY:
Although protein kinase inhibitors (PKIs) have proved effective in treating many cancers, few patients receiving PKIs may experience rare but life-threatening hepatotoxicity such as hepatic failure. Today, there is no large-scale retrospective pharmacovigilance study focusing on protein kinase inhibitors-related hepatotoxicity.

The objective was to investigate reports of hepatotoxicity related to protein kinase inhibitors using FDA Adverse Event Reporting System (FAERS).

DETAILED DESCRIPTION:
The investigators plan to include FDA approved PKIs from PKIDB, a curated, annotated and updated database of protein kinase inhibitors (https://www.icoa.fr/pkidb/).

The search terms of hepatotoxicities will be extracted from "Drug related hepatic disorders-comprehensive search (SMQ)" in MedDRA (Medical Dictionary for Regulatory Activities).

ELIGIBILITY:
Inclusion Criteria:

* Case reported in the FAERS database of individual safety case reports at the time of the extraction,
* Patients treated with at least 1 PKIs.

Exclusion Criteria:

* Chronology not compatible between the PKIs and hepatotoxicities

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cancer patients treated with protein kinase inhibitors and experiencing hepatotoxicities.
Sampling Method: Non-Probability Sample
Enrollment: 600000 (Estimated)
Dates: Start 2022-06-19 (Actual); Primary Completion 2022-07-20 (Estimated); Study Completion 2022-08-10 (Estimated)

PRIMARY OUTCOMES:
Hepatotoxicities cases reports related to PKIs (from FAERS database). | From 2004 to Sep, 2021
  The investigators plan to identify number of cases of hepatotoxicities (especially severe toxicities such as hepatic failure) reports related to PKIs reported in the FAERS database by using reporting odds ratios (ROR) and information component (IC), two common method in disproportionality analysis. Clinical features such as gender, age and indications will be displayed, too.

SECONDARY OUTCOMES:
Description of the time to onset of hepatotoxicities after PKIs exposure. | From 2004 to Sep, 2021
  The investigators plan to conduct a time to onset analysis of PKIs-related hepatotoxicities using weibull distribution
Description of the fatality cases. | From 2004 to Sep, 2021
  Fatality cases of PKIs-related hepatotocities will be described.

CONTACTS AND LOCATIONS:
Locations (1):
- Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No